CLINICAL TRIAL: NCT06869889
Title: Fluoroscopy-Guided Retrolaminar Block Versus Local Wound Infiltration for Post Lumbar Discectomy Analgesia: A Double-Blinded, Randomized Trial
Brief Title: Analgesia Following Lumbar Discectomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Spine surgeries Analgesia
Record Dates: First submitted 2025-02-25; First posted 2025-03-11 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-09

CONDITIONS: Analgesia; Disk Herniated Lumbar; Local Infiltration
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retrolaminar block group (Active Comparator): After confirming the correct position using imaging with a C-Arm device, the patient will receive a retrolaminar block on both sides at the level of the operated disc.
  Interventions: Procedure: Retrolaminar plane block
- Local Infiltration group (Active Comparator): The patient will receive local wound infiltration following the completion of the surgical steps with the patient in the prone position using a local anesthetic solution, tailored to the specific conditions surrounding the incision site.
  Interventions: Procedure: Local wound infiltration

INTERVENTIONS:
Procedure: Retrolaminar plane block — Retrolaminar plane infiltration with the local anesthetic mixture.
  Arms: Retrolaminar block group
Procedure: Local wound infiltration — Local infiltration along the surgical incision.
  Arms: Local Infiltration group

SUMMARY:
Lumbar discectomy surgeries are often the last option for patients with disc herniation who do not improve with conservative treatments. However, these procedures can lead to significant perioperative pain that may become chronic without effective management. While intravenous opioids are commonly used for pain control, they can complicate recovery and pose risks like dependence. In contrast, regional anesthetic techniques offer advantages such as quicker recovery, better postoperative pain relief, and reduced opioid use, which can lead to shorter hospital stays. Our study aims to compare the effectiveness of the retrolaminar block with local wound infiltration for pain management following posterior lumbar discectomy surgeries, potentially improving patient outcomes.

DETAILED DESCRIPTION:
Lumbar discectomy surgeries are the last resort for disc herniation patients not responding to conservative treatment. However, these surgeries are associated with annoying perioperative pain that could be severe and progress to chronic pain if not managed properly. There is no consensus regarding the best approach for postoperative pain management following spine surgeries. Intravenous opioids are still the primary agents used for perioperative pain control, which can complicate the postoperative recovery with the associated side effects and the risk of opioid dependence. Regional anesthetic techniques for spine surgeries allow rapid recovery, prolonged postoperative analgesia, and less opioid consumption, which decreases hospital stays. The current study will compare the analgesic efficacy of the retrolaminar block to the local wound infiltration following posterior lumbar discectomy surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgical decompression of single-level herniated lumbar disc.

Exclusion Criteria:

* Opioid-dependent patients.
* Known hypersensitivity to bupivacaine.
* Diabetic patients.
* Uncooperative patient or with altered mental status.
* Previous spine surgery.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2025-03-12 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of patients who required rescue analgesia | The first 24 hours postoperative.
  The percentage of patients who required rescue analgesia within the first 24 hours.
Total amount of opioid consumption | The first 24 hours postoperative.
  The total opioid consumption within the first 24 hours postoperative.

SECONDARY OUTCOMES:
The Numerical Pain Rating Scale | The first 24 hours postoperative.
  On a scale of 0-10, the patient will be asked to classify postoperative pain as the following 0: no pain, and 10: maximum imaginable pain. Postoperative pain will be assessed at 1,2,4,6,12,18, and 24 hours postoperative.
Duration of the surgical intervention. | The first 2 hours.
  Duration of surgery in minutes.
Patient satisfaction (quality of life questionnaire) | At the end of the first 24 hours postoperative.
  Patient satisfaction will be assessed using a 7-point Likert-like verbal rating scale. The patient will be asked to express their level of satisfaction 24 hours after the procedure, using the following scale: 1 = extremely dissatisfied, 2 = dissatisfied, 3 = somewhat dissatisfied, 4 = neutral, 5 = somewhat satisfied, 6 = satisfied, and 7 = extremely satisfied .

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Mohamed Nasr, MD, Study Director — Department of Anesthesia, Intensive Care & Pain Management, Zagazig University
Locations (1):
- Zagazig university hospital, Zagazig, Egypt

REFERENCES:
- [Background] Awadalla AM, Aljulayfi AS, Alrowaili AR, Souror H, Alowid F, Mahdi AMM, Hussain R, Alzahrani MM, Alsamarh AN, Alkhaldi EA, Alanazi RC. Management of Lumbar Disc Herniation: A Systematic Review. Cureus. 2023 Oct 29;15(10):e47908. doi: 10.7759/cureus.47908. eCollection 2023 Oct. PMID 38034203
- [Background] Prabhakar NK, Chadwick AL, Nwaneshiudu C, Aggarwal A, Salmasi V, Lii TR, Hah JM. Management of Postoperative Pain in Patients Following Spine Surgery: A Narrative Review. Int J Gen Med. 2022 May 2;15:4535-4549. doi: 10.2147/IJGM.S292698. eCollection 2022. PMID 35528286
- [Background] Tao T, Zhou Q. [Efficacy of erector spinae block versus retrolaminar block for postoperative analgesia following posterior lumbar surgery]. Nan Fang Yi Ke Da Xue Xue Bao. 2019 Jun 30;39(6):736-739. doi: 10.12122/j.issn.1673-4254.2019.06.17. Chinese. PMID 31270055
- [Background] Liu D, Xu X, Zhu Y, Liu X, Zhao F, Liang G, Zhu Z. Safety and Efficacy of Ultrasound-Guided Retrolaminar Block of Multiple Injections in Retroperitoneal Laparoscopic Nephrectomy: A Prospective Randomized Controlled Study. J Pain Res. 2021 Feb 5;14:333-342. doi: 10.2147/JPR.S282500. eCollection 2021. PMID 33574697